CLINICAL TRIAL: NCT07095296
Title: Effect of a Culturally Tailored Health Education Intervention Based on Social Cognitive Theory and the Theory of Planned Behavior on Postnatal Care Utilization Among Postpartum Women in Ethiopia
Brief Title: Effect of Culturally Tailored Health Education on Postnatal Care Use Among Postpartum Women in Ethiopia
Acronym: ECTHE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Responsible Party: Principal Investigator, Firew Tiyare, Principal Investigator, Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ECTHE-Ethiopia
Record Dates: First submitted 2025-07-08; First posted 2025-07-31 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Intervention
Keywords: PNC; Counseling; Health education; Newborn care; Cluster Randomized Trial
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: This study is designed as a two-arm cluster randomized controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): The control group will not receive the culturally tailored intervention. Instead, participants in this group will receive the standard routine antenatal care and postnatal health education currently provided at health facilities.
- intervention (Experimental): Women in the experimental group will receive four educational sessions, each lasting approximately 15 to 20 minutes, delivered after the completion of routine ANC services. The sessions will be conducted in small groups, with one midwife assigned to every five pregnant women, and included verbal interaction, video presentations, and practical demonstrations.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Health Education — The intervention-a culturally tailored and redesigned health education-will be guided by established behavioral theories, namely the Theory of Planned Behavior (TPB) and Social Cognitive Theory (SCT) and implemented in a culturally sensitive manner. The TPB focuses on attitudes toward utilizing PNC services, the influence of subjective norms such as cultural norm, and their perceived behavioral control including transportation (34), while SCT emphasizes self-efficacy, social modeling, and reinforcement(35). Both TPB and SCT have been extensively validated in various health behavior studies, supporting their relevance and applicability in this context(36, 37).
  Our intervention will consist of a structured training foe health extension worker and mentorship program. The intervention package, including the training curriculum and implementation manual, will be developed in accordance with guidelines from the World Health Organization (WHO) and the Federal Ministry
  Arms: intervention

SUMMARY:
This clinical study aims to find out if a redesigned health education program-one that respects local cultural beliefs and is based on well-known behavior change theories-can help improve how well mothers care for their newborns and how often they use postnatal care services. The main hypothesis is that culturally tailored health education provided by trained midwives will lead to: 1. Increased use of postnatal care services by mothers after childbirth, and 2. Improved knowledge among mothers about how to care for their newborns.

In the study, midwives will first be trained in how to provide this culturally appropriate health education. Then, the trained midwives will deliver four health education sessions-once a month-to pregnant women during their regular antenatal (before birth) visits at health facilities.

DETAILED DESCRIPTION:
Rationale and Background:

Despite the critical role of postnatal care (PNC) in reducing neonatal morbidity and mortality, it remains one of the least utilized maternal health services in Ethiopia. According to national surveys, only 35% of newborns receive a PNC checkup within the first three days postpartum. Cultural beliefs such as postpartum seclusion, fears of exposure to the "evil eye", lack of awareness, and economic barriers contribute significantly to low uptake.

Midwives serve as the primary providers of perinatal care but often lack the necessary tools, training, and culturally sensitive materials to communicate effectively. Existing counseling practices are generic, inadequately address local beliefs, and often fail to promote sustained behavior change. Thus, this study seeks to address these gaps.

The current study is a cluster-randomized controlled trial designed to evaluate the effectiveness of a culturally tailored health education intervention in improving postnatal care (PNC) utilization and maternal knowledge of newborn care among postpartum women in the Jimma Zone of Ethiopia. The intervention is grounded in two well-established behavior change models: Social Cognitive Theory and the Theory of Planned Behavior, and will be adapted to the local context through formative research, expert validation, and pilot testing.

The study targets two primary objectives:

1. To assess the effect of culturally tailored training for midwives on postnatal care (PNC) service utilization among postpartum women.
2. To evaluate whether the intervention improves maternal knowledge of newborn care practices.

Intervention Overview:

The intervention consists of a structured health-education training program for midwives and health extension workers, with a focus on culturally tailored postnatal health education. Following the training, the health extension workers-under the supervision of midwives-will deliver four educational sessions to pregnant mothers' forums on a monthly basis. The session content is aligned with WHO and Ethiopian Federal Ministry of Health guidelines and is informed by the Social Cognitive Theory (SCT) and the Theory of Planned Behavior (TPB). Each session lasts approximately 10 to 20 minutes.

Each session has a specific focus:

Session 1: Value clarification, barriers to care, and goal-setting. Session 2: Benefits of PNC and consequences of missed care (role modeling and video demonstrations).

Session 3: Essential newborn care topics (e.g., danger signs, hygiene, cord care).

Session 4: Summary and self-evaluation through peer group discussions.

Sample size:

The study is powered to detect a 20% increase in PNC use relative to an expected rate of 28% in the control group. The sample size was determined using the Hayes and Bennett formula for cluster-randomized trials comparing two proportions. The investigators assumed a primary outcome of postnatal care (PNC) visit completion with a baseline proportion of 28%, and expected an improvement of 20% points in the intervention group.

With an average of 20 mothers per cluster, a 2:1 control-to-intervention allocation ratio, and ICC of 0.10, the investigators need to 14 treatment and 28 control clusters, with a total final sample size of N=820 to achieve power 0.9. the investigators will enroll an additional 3 mothers (15%) in each cluster to allow for some attritions).

Sampling procedure:

A multistage sampling approach using Probability Proportional to Size (PPS) will be employed to identify study participants. In the first stage, woredas will be selected using PPS based on their population size. In the second stage, two health facilities will be randomly selected from each sampled woreda. From the selected facilities, the catchment kebeles will be stratified by study arm, after which one kebele will be selected from the intervention arm and two kebeles from the control arm using simple random sampling. In the final stage, a fixed sample of 23 eligible mothers will be randomly selected from each selected kebele using household lists or community registers. This systematic and weighted sampling process ensures representativeness across woredas, facilities, and kebeles while maintaining balance between study arms.

Data Collection:

Baseline data will be collected through face-to-face interviews at enrollment using structured questionnaires on tablets (KoboToolbox). Endline data will be collected via telephone, or in-person home visits for unreachable participants. Data collection will be carried out by trained Master of Public Health (MPH) students blinded to treatment allocation.

Primary and Secondary Outcomes:

The primary outcomes of the study is postnatal care (PNC) utilization, while secondary outcomes newborn care knowledge. PNC utilization is defined according to the World Health Organization (WHO) recommendations, that postnatal care (PNC) should be provided through at least four scheduled contacts; first postnatal visit should occur within 24 hours of birth, followed by subsequent visits on Day 3 (48-72 hours), between Days 7-14, and at six weeks postpartum. Newborn care knowledge among mothers will be categorized as "good knowledge" or "poor knowledge", with the cutoff set at mothers correctly answering at least 50% of the items on the maternal knowledge of newborn care questionnaire. The covariates in this study includes sociodemographic, economic status, distance from health facility, and household decision making.

Statistical Analysis:

Analyses will follow the intention-to-treat principle. For binary outcomes (PNC use, knowledge level), generalized linear models (e.g., logistic regression) with standard errors clustered at the facility level will be used. Both adjusted and unadjusted models will be reported, adjusting for potential residual confounders including education and parity. Sensitivity analyses will account for missing data using multiple imputation if appropriate.

Compliance:

To ensure compliance during the intervention study, the investigators will consider flexible scheduling to accommodate mothers' availability. Monitoring and follow-ups will be used to help track implementation and presence of the trained Midwives throughout the study. Contact details will be collected at enrollment, and reminder phone calls or messages will be sent to mothers to encourage participation.

Strategies to minimize confounder and bias:

Given the random assignment of treatments, confounding is not expected to be a major concern. However, to account for potential residual confounding, the investigators will adjust for education level and number of previous pregnancies in the regression model. To minimize spillover effects, randomization will be conducted at the health facility level. Additionally, to reduce observer bias, data collectors will be blinded to group allocation.

Quality Assurance:

The study includes a comprehensive quality assurance plan:

* Pretested instruments and SOPs for recruitment, data collection, and intervention delivery.
* Regular field supervision, debriefings, and fidelity checks.
* Embedded data validation rules in the electronic platform.
* Source data verification on a sample basis using facility records and maternal cards.

An audit trail and detailed logbook (digital and paper-based) will capture day-to-day activities and data issues. All research staff will be trained in ethics, confidentiality, and SOP adherence prior to study initiation.

Data management plan:

This research project will implement a comprehensive Data Management Plan (DMP) to ensure the responsible handling, preservation, and accessibility of all research data generated. All raw and processed data will be systematically collected, documented, and stored in secure, access-controlled repositories in compliance with Swiss TPH guidelines. Metadata will be standardized following the FAIR (Findable, Accessible, Interoperable, and Reusable) data principles to facilitate future reuse and reproducibility. To prevent data loss due to hardware failure or human error, regular backups will be performed using both local and cloud-based storage solutions.

An audit trail will be maintained throughout the project to document all modifications made to the data-clearly recording when, how, and by whom changes were made-thereby enhancing transparency and reproducibility. A comprehensive data dictionary will accompany all datasets, providing clear definitions of variables, coding schemes, and units of measurement to ensure consistency across collaborators and future users. Data cleaning procedures will be conducted in Stata and fully documented using well-annotated do-files. Additionally, a logbook will be maintained in both digital and physical formats, as appropriate, to capture day-to-day research activities, data issues encountered, decisions made, and updates to protocols-further supporting the audit trail and ensuring full traceability of the research process.

Ethical Oversight:

The study will receive ethical approval from the Institutional Review Board of Jimma University and the Ethics Committee of Northwest and Central Switzerland (EKNZ), with local approvals from regional health bureaus. Written informed consent will be obtained from all participants. Illiterate participants will be consented in the presence of a non-research witness.

Confidentiality will be maintained through de-identified data and secure storage protocols. Data will be retained for a maximum of 20 years at Swiss TPH and Jimma University, in accordance with institutional policy.

Participants will not receive financial incentives. Participation will be voluntary, with the right to withdraw at any point without consequence.

ELIGIBILITY:
Cluster-Level Eligibility Criteria:

To be eligible for inclusion, clusters must meet the following criteria:

* A catchment population size of at least 5,000 people
* An average of more than 50 antenatal care (ANC) visits per month
* Location in a peri-urban area to facilitate participant follow-up

Individual-Level Eligibility Criteria (for mothers):

* Gestational age between 20 and 24 weeks at the time of enrollment
* Residence within one hour's travel distance from the selected health facility

Individual-Level Exclusion Criteria:

* Mothers who plan to relocate from the selected cluster area before or shortly after delivery
* Mothers who do not speak either Afan Oromo or Amharic, as these are the languages used for delivering the intervention.
* Mothers who have already completed all recommended postnatal care visits during their most recent previous birth

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnancy
Enrollment: 864 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Postnatal care use | From birth to the end of postnatal period(6th week)
  PNC utilization will be assessed based on the World Health Organization (WHO) recommendations, which define adequate postnatal care as having four scheduled contacts: within 24 hours of birth, on Day 3 (48-72 hours), between Days 7-14, and at six weeks postpartum.
  Data will be collected using a structured maternal postnatal care follow-up questionnaire administered during endline interviews. This questionnaire includes items capturing self-reported timing and number of PNC visits, supplemented by verification from clinic records where available.
  For the primary analysis, PNC utilization will be coded as a binary variable: 1 (Yes) - if the mother attended at least two postnatal care visits and 0 (No) - if the mother attended fewer than two visits. This threshold reflects a more feasible level of access in the study setting.
  For the secondary analysis, attendance of all four WHO-recommended visits will be assessed as an indicator of higher adherence to WHO standards.

SECONDARY OUTCOMES:
Newborn care knowledge | From birth to the end of fourth week
  Maternal knowledge of newborn care will be assessed using a structured questionnaire titled the "Maternal Knowledge of Newborn Care Questionnaire", developed based on World Health Organization (WHO) guidelines and existing validated tools.
  The consists of 16 items grouped into key dimensions of essential newborn care, including breastfeeding, recognition of neonatal danger signs, vaccination, hygiene practices, cord and eye care, and sunlight exposure. Each correct response will be scored as 1, and incorrect or "don't know" responses as 0. The questionnaire has a total score ranging from 0 to 22, where 22 indicates the highest level of knowledge and 0 represents no correct knowledge.
  Mothers will be categorized as follows: Good knowledge - correctly answering at least 50% of the items and Poor knowledge - correctly answering less than 50% of the items. This binary classification will serve as the primary metric for evaluating newborn care knowledge in the analysis.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This decision is based on the need to protect participant privacy and confidentiality, as the dataset contains sensitive health information that cannot be fully de-identified without compromising data integrity. Additionally, the consent form and ethical approval for this study do not include provisions for public sharing of raw participant-level data. Summary results, however, will be shared in line with WHO and ClinicalTrials.gov requirements.